CLINICAL TRIAL: NCT03314506
Title: Adipose Tissue Cellular Response to Exercise in Healthy Humans
Acronym: FLOW
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Michigan (Other)
Responsible Party: Principal Investigator, Jeffrey F Horowitz, Associate Professor, Movement Science, School of Kinesiology, University of Michigan
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: HUM00131070
Record Dates: First submitted 2017-09-27; First posted 2017-10-19 (Actual); Last update posted 2022-03-21 (Actual); Status verified 2022-03

CONDITIONS: Metabolic Disease; Adipose Tissue
Keywords: exercise
MeSH Terms: conditions — Metabolic Diseases; Motor Activity | interventions — Exercise

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Trial (Experimental): Subjects will need to come to the Substrate Metabolism Laboratory in the morning around 7:00 AM. After about a 15-30 minute rest, the study team will collect a blood sample from the subject's hand or forearm. The study team will also obtain a small sample of fat tissue from the area just underneath the skin near the belly button. Next, subjects will exercise on a treadmill at a moderate intensity for about 1 hour. Immediately after exercising the study team will collect a blood sample. The subject will remain resting in the laboratory for 3 hours after exercise, and then the study team will collect another blood and fat tissue sample. Upon completion, the subject will be provided a snack before leaving the laboratory.
  Interventions: Other: Exercise

INTERVENTIONS:
Other: Exercise — Subjects will exercise on a treadmill for 1 hour at a moderate intensity (approximately 70% of their predicted VO2peak).

SUMMARY:
The purpose of this study is to measure the effects of a single session of exercise on changes in the cellular composition of the body fat of humans.

DETAILED DESCRIPTION:
Fat tissue is far more than just a place where humans store body fat. Fat tissue contains many different types of cells, such as immune cells, endothelial cells, and fat precursor cells. Differences or changes in the number of immune cells, endothelial cells, and fat precursor cells in fat tissue can have a great impact on metabolic health. The abundance of all immune cells, endothelial cells, and fat precursor cell types are known to change when a person loses or gains weight. For example, the abundance of inflammatory cells is often found to decrease markedly with weight loss - and this change has been linked to the profound improvements in metabolic health that occur with weight loss. In contrast, the effects of exercise on immune cells, endothelial cells, and fat precursor cells in fat tissue is not known. Determining the effects of exercise on changes in the cellular composition within fat tissue will provide important information for optimizing lifestyle interventions aimed at improving metabolic health.

ELIGIBILITY:
Inclusion Criteria:

* Age: 18-40
* Body Mass Index: 20-27 kg/m2
* Regular exercise (less than or equal to 3 days/week of aerobic exercise; 30-60 minutes/session at moderate and vigorous intensities)
* Women must have regularly occurring menses and must be premenopausal

Exclusion Criteria:

* Blood pressure greater than 140/90 mm Hg
* Pregnant or lactating
* Evidence/history of cardiovascular or metabolic disease
* Medications known to affect lipid or glucose metabolism, or inflammation

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2017-11-01 (Actual); Primary Completion 2019-08-08 (Actual); Study Completion 2019-08-08 (Actual)

PRIMARY OUTCOMES:
Quantifying the change in markers of macrophage abundance in adipose tissue | 1 day
  The stromovascular fraction will be isolated from subcutaneous lipo-aspirate samples by collagenase digestion and a series of filtration/wash steps (routinely performed by our lab). This isolation protocol has been optimized to yield the minimum number of stromal cells required to identify and recover the following cell populations by fluorescence-activated cell sorting (FACS), listed as cell surface stain = cell type: CD64+/CD11c+ = macrophages
  FACS will be performed at the University of Michigan Flow Cytometry Core, and sorted cells will be recovered for subsequent gene expression analysis using the StepOnePlus real time PCR system (Life Technologies) with fluorescent probe-based assays.

SECONDARY OUTCOMES:
Quantifying the change in markers of endothelial cell and pre-adipocytes in adipose tissue | 1 day
  The stromovascular fraction will be isolated from subcutaneous lipo-aspirate samples by collagenase digestion and a series of filtration/wash steps (routinely performed by our lab). This isolation protocol has been optimized to yield the minimum number of stromal cells required to identify and recover the following cell populations by fluorescence-activated cell sorting (FACS), listed as cell surface stain = cell type: CD34+/CD31+ = endothelial cells
  FACS will be performed at the University of Michigan Flow Cytometry Core, and sorted cells will be recovered for subsequent gene expression analysis using the StepOnePlus real time PCR system (Life Technologies) with fluorescent probe-based assays.

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey F Horowitz, Principal Investigator — University of Michigan
Locations (1):
- University of Michigan, Ann Arbor, Michigan, United States